CLINICAL TRIAL: NCT00670774
Title: A Single Center, Open-label Study to Determine the Safety and Efficacy of a Dosing Regimen of Eculizumab Added to Conventional Treatment in the Prevention of Antibody-mediated Rejection (AMR) in Positive Crossmatch Living Donor Kidney Transplantation
Brief Title: Dosing Regimen of Eculizumab Added to Conventional Treatment in Positive Cross Match Living Donor Kidney Transplant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mark Stegall (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Mark Stegall, MD, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-007208
Record Dates: First submitted 2008-04-28; First posted 2008-05-02 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-05

CONDITIONS: Kidney Transplant
Keywords: Kidney; Transplant; donor
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eculizumab (Experimental): Patients received eculizumab intravenously according to details provided in the intervention description.
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — * Patients will be given 1200 mg of eculizumab intravenously over 30 minutes, 1 hour prior to surgery.
  * Patients will be given 900 mg of eculizumab on Day 1 post-transplant.
  * Patients will then be given 900 mg of eculizumab weekly through 4 weeks post-transplant
  * At week 4, patients will be assessed for B cell flow cytometry cross match (FCXM). Patients with B cell FCXM less than 200 will stop eculizumab treatment. Patients with B cell FCXM greater than or equal to 200 will continue eculizumab treatment every 14 days from week 5 through week 9. The dose will be increased to 1200 mg and dosing will now be every 2 weeks instead of weekly. Similar "discontinuation assessments" will be performed at week 9, 26, 39 and 52.
  * In addition, eculizumab 600 mg will be administered immediately after each plasmapheresis (PP) and immediately after any fresh frozen plasma (FFP) that is given post-transplant during the treatment period
  Other Names: Soliris

SUMMARY:
A strongly positive crossmatch has long been considered an absolute contraindication to kidney transplantation and most patients with anti-human leukocyte antigen (HLA) antibody never were able to receive a kidney transplant. Over the past decade, significant progress has been made in overcoming early antibody-mediated renal allograft injury. Our group has performed more than 200 such transplants providing the possibility of transplant to previously untransplantable patients. Despite our best efforts, transplantation in these patients is still complicated by a high rate of acute humoral rejection (AHR).

Patients included in this study will be those who have demonstrable anti-HLA antibody specific for their living donor. It is our hypothesis that blockade of terminal complement activation at the time of transplant in combination with our current protocols will reduce the incidence of AHR in patients with anti-donor HLA antibody.

DETAILED DESCRIPTION:
The eculizumab dosing regimen was modified from that used in the treatment of paroxysmal nocturnal hemoglobinuria and consisted of 1200 mg immediately prior to transplantation, 600 mg on postoperative day 1, and 600 mg weekly thereafter for 4 weeks. At week 4, assessment of DSA levels was performed. Eculizumab was discontinued in patients whose DSA had significantly decreased (B flow crossmatch channel shift<200). In patients with persistently high DSA and thus believed to have continued high risk for AMR, eculizumab treatment continued (1200 mg week 5, and then every 2 weeks). Another DSA assessment was performed at week 9 and eculizumab was discontinued if the B flow crossmatch channel shift was <200.

The eculizumab group were compared to a historical control group consisting of consecutive transplants between 1/1/2005 and 1/10/2017 who met the inclusion criteria. The historical control group had been treated with a similar plasma exchange based protocol without eculizumab.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age
2. Has end stage renal disease (ESRD) and is to receive a kidney transplant from a living donor (LD) to whom he/she has either:

   1. A positive crossmatch requiring pretransplant desensitization (defined as a positive T-cell FCXM of greater than or equal to 300 but less than 450 prior to desensitization, or as a positive B-cell FCXM of > 300 but < 450 prior to desensitization with demonstrable Class II donor specific alloantibody (DSA) on solid-phase assays). Subsequent to desensitization, patient must have, at the time of transplant, a T-cell and B-cell FCXM less than 300; or
   2. A positive crossmatch not requiring desensitization (defined as FCXM between 200 and 299)
3. Willing to comply with the protocol
4. Females of child-bearing potential must have a negative pregnancy test (serum β-HCG) and sexually active females must agree to use a reliable and medically approved method of contraception
5. Willing and able to give written informed consent
6. Vaccinated against Neisseria meningitides (quadrivalent vaccine), Pneumococcus or H. influenzae at least two weeks prior to beginning desensitization

Exclusion Criteria:

1. Unstable cardiovascular condition
2. Previous splenectomy
3. Active bacterial or other infection which is clinically significant in the opinion of the investigator
4. Known or suspected hereditary complement deficiency
5. Participation in any other investigational drug study or was exposed to an investigational drug or device within 30 days of randomization
6. Pregnant, breast-feeding, or intending to conceive during the course of the study, including the two month follow-up period after drug discontinuation
7. Known hypersensitivity to the treatment drug or any of its excipients
8. History of illicit drug use or alcohol abuse within the previous year
9. History of meningococcal disease
10. Medical condition that, in the opinion of the investigator, might interfere with the patient's participation in the study, pose an added risk for the patient, or confound the assessment of the patient (e.g. severe cardiovascular or pulmonary disease)
11. Previously been enrolled in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Stegall, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Stegall MD, Diwan T, Raghavaiah S, Cornell LD, Burns J, Dean PG, Cosio FG, Gandhi MJ, Kremers W, Gloor JM. Terminal complement inhibition decreases antibody-mediated rejection in sensitized renal transplant recipients. Am J Transplant. 2011 Nov;11(11):2405-13. doi: 10.1111/j.1600-6143.2011.03757.x. Epub 2011 Sep 22. PMID 21942930
- [Derived] Bentall A, Tyan DB, Sequeira F, Everly MJ, Gandhi MJ, Cornell LD, Li H, Henderson NA, Raghavaiah S, Winters JL, Dean PG, Stegall MD. Antibody-mediated rejection despite inhibition of terminal complement. Transpl Int. 2014 Dec;27(12):1235-43. doi: 10.1111/tri.12396. Epub 2014 Aug 20. PMID 24990476

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive kidney transplant patients recruited between 1/6/2008 and 1/8/2010 were recruited at Mayo Clinic in Rochester, Minnesota.
Pre-assignment Details: 31 subjects signed informed consent, but 5 patients were screen failures and did not start the study.
Period: Overall Study
Arm/Group | Eculizumab
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Only subjects who received eculizumab and were transplanted were included in the baseline characteristics.
Arm/Group | Eculizumab
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian white | 24
  Hispanic | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26
Donor Specific Alloantibody [Mean (Standard Deviation); unit: MCF shift from NC] — The presence and amount of donor specific alloantibody (DSA) was assessed using cell-based T- and B-flow cytometric crossmatch channel shift. The channel shift is the observed number of channels (raw fluorescence) above the negative control. The units for DSA are mean channel fluorescence (MCF) shifts from negative control (MCF shift from NC).
  MCF shift from NC | 330 (84)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Antibody-Mediated Rejection (AMR) in the First 3 Months After Living Donor Kidney Transplantation
Description: AMR can cause acute graft loss or shorten allograft survival. Renal allograft biopsies were obtained percutaneously using ultrasound guidance processed for light microscopy and immunofluorescence for peritubular capillary staining for C4d. All biopsies were reviewed by a pathologist in a blinded fashion. AMR was diagnosed using standard Banff criteria in combination with graft dysfunction (increase in serum creatinine >/=0.3 mg/dL over nadir.)
Time Frame: up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 26
Participants | 2

2. Secondary Outcome: Number of Patients Developing High DSA Levels at Less Than or Equal to 3 Months
Description: High DSA levels were defined as B flow cross match channel shift >350 at any time point in the first 3 months.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 26
Participants | 13

3. Secondary Outcome: Number of Patients Requiring Splenectomy
Description: A splenectomy is a surgical operation involving removal of the spleen. Splenectomy was performed for severe AMR in the setting of a rising serum creatinine (usually >2.0) and a rising serum DSA level despite daily plasma exchange treatments.
Time Frame: 1 year
Population: 10 subjects discontinued early (<1 year) according to protocol because they had a B flow cytometric crossmatch (BFMX) <200.
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 16
Participants | 0

4. Secondary Outcome: Graft Dysfunction in First Month Post Transplant
Description: (Maximum serum creatinine-nadir serum creatinine)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Eculizumab
Number analyzed (Participants) | 26
mg/dL | 0.45 (0.37)

5. Secondary Outcome: Length of Follow-up
Description: Following the completion of dosing, subjects were to return for follow-up visits at 3 and 6 months post transplant to obtain biopsies and collect follow-up data. Subjects who continued the drug for 12 months were to receive their final assessment at 15 months.
Time Frame: up to 15 months
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Eculizumab
Number analyzed (Participants) | 26
months | 11.9 (6.1)

6. Secondary Outcome: Number of Subjects With Graft Survival at One Year
Description: Graft survival means the kidney has not been rejected by the body.
Time Frame: 1 year
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 16
Participants | 16

7. Secondary Outcome: Number of Subjects Receiving Posttransplant Plasma Exchange (PE)
Description: Plasma exchange is needed when there is poor kidney functioning, and donor specific alloantibody (DSA) is high
Time Frame: up to one year
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 26
Participants | 3

8. Secondary Outcome: Transplant Glomerulopathy Incidence at One Year
Description: Transplant glomerulopathy is a morphologic lesion of renal allografts that is characterized histologically by duplication and/or multilayering of the glomerular basement membrane. It is widely accepted as a manifestation of chronic antibody-mediated rejection (AMR). This is determined by histology.
Time Frame: 1 year
Population: 10 subjects discontinued early (<1 year) according to protocol because they had a B flow cytometric crossmatch (BFMX) <200. An additional subject did not have a biopsy done at one year.
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 15
Participants | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Eculizumab
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 26/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=26)
Elevated Creatinine (Renal and urinary disorders) | 2 (2)
Cross-connection end-to-end of the segments of the same ureter (Renal and urinary disorders) | 1 (1)
Swelling and erythema of left hand (Skin and subcutaneous tissue disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 4 (4)
Diarrhea and vomiting (Gastrointestinal disorders) | 3 (3)
Rapid pulse (Cardiac disorders) | 1 (1)
Acute dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dissection of the iliac (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2
Headache (General disorders) | 1 (1)
Hypercalcemia (General disorders) | 1 (1)
Tonic-colonic seizure (General disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Tertiary Hyperparathyroidism (General disorders) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Small bowel perforation (Injury, poisoning and procedural complications) | 1 (1)
Elevated Creatinine (Renal and urinary disorders) | 1 (1)
Hyperkalemia (Renal and urinary disorders) | 2 (2)
Wound dehiscence (General disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1)
Pain following kidney biopsy (Renal and urinary disorders) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Acute humoral rejection (Renal and urinary disorders) | 1 (1)
Ulnar fracture secondary to a dog bite (Injury, poisoning and procedural complications) | 1 (1)
Lymphocele (Blood and lymphatic system disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Pulmonary blastomycosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Abdominal pain secondary to constipation (Gastrointestinal disorders) | 1 (1)
Bleeding following kidney biopsy (Renal and urinary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Light headed (General disorders) | 1 (1)
Diaphoresis (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-03-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT00670774/Prot_SAP_000.pdf